CLINICAL TRIAL: NCT05268172
Title: Single-arm Open Multicenter Study of IFN-γ Combined With T Cells in the Treatment of Refractory Malignant Pleural Effusion Tumors
Brief Title: IFN-γ Combined With T Cells in the Treatment of Refractory Malignant Pleural Effusion and Ascites
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Affiliated Hospital of Jiangnan University (Other)
Collaborators: Sichuan University (Other); Zhejiang Provincial People's Hospital (Other); Hunan Cancer Hospital (Other); West China Hospital (Other); Wuxi People's Hospital (Other); Shenzhen Second People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1362566548
Record Dates: First submitted 2021-12-06; First posted 2022-03-07 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Pleural Effusion, Malignant
MeSH Terms: conditions — Pleural Effusion, Malignant | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IFN- Y combined with T cells (Experimental): First, IFN-γ was combined with CIK cells. After three failed treatments, the CIK cells were replaced with T cells. After three failed treatments, CART cells were finally replaced.
  Interventions: Drug: IFN-γ and CIK cells, Tcm cells or CAR T cells

INTERVENTIONS:
Drug: IFN-γ and CIK cells, Tcm cells or CAR T cells — A 50ng/ mL IFN-γ solution was prepared, and the required volume of IFN-γ solution was calculated according to the final concentration of 5ng/ mL according to the volume of pleural fluid or ascites of the patient. CIK cells were injected 1.0-2.0×109 on the second day and review three days later.T cells and CAR T cells were selected sequentially according to the re-examination of pleural fluid or ascites.

SUMMARY:
The purpose of this study was to evaluate the efficacy of IFN- Y combined with T cells in the treatment of refractory malignant pleural effusion and acties, using a multicenter, single-arm, open design.

DETAILED DESCRIPTION:
Malignant pleural effusion is a common complication of malignant tumor, which usually indicates that the patient has reached the advanced stage, and about 30-40% of the patients are stubborn and refractory cases. The lack of standard therapeutic drugs and protocols in clinical practice seriously affects the anti-tumor treatment effect, quality of life and survival time of patients, and the prognosis is poor. IFN-γ can significantly induce the high expression of the costimulatory molecule ICAM-1 on tumor cells, thereby enhancing the killing of TUMOR cells by T cells. Moreover, IFN-γ can enhance the activity of CAR T cells in the presence of PD-L1-PD-1 pathway, and significantly improve the therapeutic effect of T cells on solid tumors. IFN-γ is an approved clinical treatment with known side effects and well-established symptomatic treatment. Although CIK is not a clinically approved drug, it has been used on a large scale in China with good safety and has entered the medical insurance of some provinces and cities. Tcm is an improved CIK cell and has good safety. Many clinical studies have been carried out, and no serious toxic and side effects have been observed.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients: ≥18 years old;
2. Gastric cancer, colon cancer, lung cancer, lymphoma and other tumors confirmed by histology or cytology. The guidelines recommend entry to clinical trials in accordance with the standard treatment progression recommended by each disease guideline;
3. According to iRECIST criteria, the patient should have at least one target lesion with measurable diameter line (tumor lesion CT scan length ≥10 mm, lymph node lesion CT scan short diameter ≥15 mm, scan thickness ≥ 5 mm); Or an unevaluable lesion, including but not limited to pleural effusion, bone metastasis, etc;
4. ECOG physical condition score: 0-3;
5. Estimated survival ≥3 months;
6. Good function of major organs, that is, relevant examination indexes within the first 14 days of randomization meet the following requirements:(1)Routine blood test: 1)Hemoglobin ≥ 90 g/L (no blood transfusion within 14 days); 2)Neutrophil count > 1.5×109/L; 3)Platelet count ≥ 90×109/L; (2)Biochemical examination: 1)Total bilirubin ≤ 1.5×ULN (upper limit of normal value); 2)Serum alanine aminotransferase (ALT) or AST ≤ 2.5×ULN; ALT or AST ≤ 5×ULN if liver metastasis was present; 3)Endogenous creatinine clearance ≥ 60 mL /min (Cockcroft-Gault formula); (3)Cardiac Doppler ultrasound assessment: left ventricular ejection fraction (LVEF) ≥ 50%;
7. Signed informed consent;
8. Good compliance, family members agreed to cooperate with survival follow-up.

Exclusion Criteria:

1. Participated in clinical trials of other drugs within four weeks;
2. Patients have a history of other tumors, except cervical carcinoma in situ, treated squamous cell carcinoma or bladder epithelial tumor (Ta and TIS), or other malignant tumors that have received radical treatment (at least 5 years prior to enrollment);
3. Patients with cardiac clinical symptoms or diseases that are not well controlled, such as NYHA grade 2 or above heart failure, unstable angina pectoris, myocardial infarction within 1 year, and clinically significant ventricular or ventricular arrhythmias requiring treatment or intervention；
4. For female subjects: surgically sterilized, postmenopausal, or have agreed to use a medically approved contraceptive during study treatment and for 6 months after the study treatment period; Serum or urine pregnancy tests must be negative during the 7 days prior to study enrollment and must be non-lactation. Male subjects: patients who are surgically sterilized or who have agreed to use a medically approved contraceptive during and for 6 months after the study treatment period；
5. Patients with active tuberculosis, bacterial or fungal infection (grade ≥2 of NCI-CTC, 3rd edition); Have HIV infection, HBV infection, HCV infection；
6. Those who have a history of psychotropic drug abuse and cannot get rid of it or have mental disorders;
7. The subject has any active autoimmune disease or a history of autoimmune disease (e.g., but not limited to: interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, nephritis, hyperthyroidism, hypothyroidism); Subjects with vitiligo or asthma in complete remission during childhood without any intervention as adults could be included; Subjects with asthma requiring medical intervention with bronchodilators were excluded)；
8. According to the judgment of the researcher, there are serious concomitant diseases that endanger the patient's safety or affect the patient's ability to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Puncture-free Survival (PuFS) | Focusing on the time from the end of the T Cells treatment procedure to the next required drainage or death
  Puncture-free Survival (PuFS) is a clinical endpoint used to measure the time duration during which a patient with a condition like malignant ascites or malignant pleural effusion remains free from needing a puncture procedure

SECONDARY OUTCOMES:
Disease control rate | The tumor shrinks or stabilizes for a certain period of time，Lasts at least 4 weeks
  Proportion of patients who had a best response rating of complete response, partial response, or stable disease
Objective response rate | 8 weeks
  Total response and partial response ratio
Molecular markers for efficacy prediction | 8 weeks
  Prediction effect
Overall survival | From the time of diagnosis of tumor to death from any cause，From initiation of study treatment until date of death from any cause, up to 100 months
  The last follow-up time of the lost patient; Patients who were still alive at the end of the study were at the end of follow-up
Progression-free survival | From time of treatment to time of disease progression or death from any cause as assessed by the investigator at each treatment period
  From time of treatment to time of disease progression or death

CONTACTS AND LOCATIONS:
Overall Officials: quan liu, doctor, Principal Investigator — Affiliated Hospital of Jiangnan University; liu quan, doctor, Study Director — Affiliated Hospital of Jiangnan University
Locations (1):
- Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
The associated efficacy is uncertain